CLINICAL TRIAL: NCT00000816
Title: Gradual Initiation of Trimethoprim/Sulfamethoxazole as Primary Pneumocystis Carinii Pneumonia Prophylaxis
Brief Title: Gradual Initiation of Sulfamethoxazole/Trimethoprim as Primary Pneumocystis Carinii Pneumonia Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 268; 11244 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Sulfamethoxazole-Trimethoprim
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: Sulfamethoxazole-Trimethoprim

SUMMARY:
To determine whether gradual initiation of sulfamethoxazole/trimethoprim (SMX/TMP) reduces the incidence of treatment-limiting adverse reactions compared to the routine initiation of the drugs for Pneumocystis carinii pneumonia (PCP) prophylaxis in HIV-infected patients.

Although a number of clinical trials have demonstrated the superiority of SMX/TMP for PCP prophylaxis, the incidence of adverse reactions to this medication is high. In a pilot study in which patients were initiated with SMX/TMP prophylaxis by gradually increasing the dose over 2 weeks, no significant adverse reactions have occurred.

DETAILED DESCRIPTION:
Although a number of clinical trials have demonstrated the superiority of SMX/TMP for PCP prophylaxis, the incidence of adverse reactions to this medication is high. In a pilot study in which patients were initiated with SMX/TMP prophylaxis by gradually increasing the dose over 2 weeks, no significant adverse reactions have occurred.

Patients are randomized to receive either gradually increasing doses of SMX/TMP suspension or routine daily initiation of SMX/TMP double strength (DS) tablets for 2 weeks. All patients will then be switched over to receive open-label SMX/TMP DS tablets daily for 10 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed if clinically indicated:

* Recombinant erythropoietin (rEPO) and G-CSF.

Allowed for symptomatic treatment of mild study drug toxicity:

* Antipyretics and analgesics (ibuprofen).
* Antihistamines (diphenhydramine HCl).
* Terfenadine or astemizole (but not allowed with concomitant antifungal or macrolide use).
* Systemic steroids.

Patients must have:

* HIV infection.
* CD4 count <= 250 cells/mm3 OR history or presence of thrush.
* No history of confirmed or probable pneumocystosis.

NOTE:

* Pregnant women are not excluded, but safety issues should be discussed with patient prior to enrollment.
* This study is appropriate for prisoner participation.
* Coenrollment in ongoing ACTG antiretroviral studies is permitted provided no new study drugs are added to the patient's drug regimen for 4 weeks before or after initiation of SMX/TMP.

Prior Medication:

Allowed:

* Prior aerosolized pentamidine and dapsone for primary PCP prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known adverse reactions to sulfa, trimethoprim, or SMX/TMP.
* Inability to comply with dosing schedule or complete dosing record.

Concurrent Medication:

Excluded:

* Procysteine.
* Glutathione.
* N-acetylcysteine (NAC).
* Antihistamines (unless used for symptomatic treatment of study drug toxicity).
* Systemic corticosteroids (unless used for replacement purposes).
* Leucovorin calcium (unless used for symptomatic treatment of study drug toxicity).
* TMP or sulfa drugs outside of the study.

Prior Medication:

Excluded at any time:

* Prior SMX/TMP as primary PCP prophylaxis.

Excluded within 4 weeks prior to study entry:

* Initiation of antiretroviral agents.
* Initiation of anti-infective agents (including SMX/TMP for another indication).

Excluded within 2 weeks prior to study entry:

* Antihistamines.
* Procysteine.
* Glutathione.
* N-acetylcysteine (NAC).
* Systemic corticosteroids (unless used for replacement purposes).
* Leucovorin calcium.
* TMP and sulfa drugs separately.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Para MF, Study Chair; Dohn MN, Study Chair; Frame P, Study Chair
Locations (42):
- United States (40):
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Para MF, Dohn M, Frame P, Becker S, Finkelstein D, Walawander A. ACTG 268 trial - gradual initiation of trimethoprim/sulfamethoxazole (T/S) as primary prophylaxis for Pneumocystis carinii pneumonia (PCP). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:65 (abstract no 2)
- [Background] Para MF, Finkelstein D, Becker S, Dohn M, Walawander A, Black JR. Reduced toxicity with gradual initiation of trimethoprim-sulfamethoxazole as primary prophylaxis for Pneumocystis carinii pneumonia: AIDS Clinical Trials Group 268. J Acquir Immune Defic Syndr. 2000 Aug 1;24(4):337-43. doi: 10.1097/00126334-200008010-00007. PMID 11015150